CLINICAL TRIAL: NCT02749487
Title: Neutrophil Lymphocyte and Platelet Lymphocyte Ratios as Predictors of Outcome in Traumatic Critically Ill Patients
Brief Title: Neutrophil Lymphocyte Ratio as a Predictor of Outcome in Critically Traumatic Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and critical care Medicine, Assiut University
Other Study IDs: IRB00009905
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Critical Care
Keywords: Critical Care; Neutrophils; Lymphocytes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cured (c): Neutrophil Lymphocyte and platelet lymphocyte ratios as Predictors of Outcome in Traumatic Critically ill Patients
  Interventions: Other: Neutrophil Lymphocyte Ratio
- Died ( M): Neutrophil Lymphocyte and platelet lymphocyte ratios as Predictors of Outcome in Traumatic Critically ill Patients
  Interventions: Other: Neutrophil Lymphocyte Ratio

INTERVENTIONS:
Other: Neutrophil Lymphocyte Ratio — Neutrophil:lymphocyte ratio (NLR) is an emerging biomarker that is used to predict mortality and morbidity. The association of this biomarker with systemic illness and its usefulness in risk assessment of critically ill patients has not been fully elucidated.

SUMMARY:
Neutrophil lymphocyte ratio NLR is an important index that evaluate the inflammatory status . It is a cost effective and readily available , and simply calculated , so that why investigators try to use it as a predictor of short term survival in the critically ill patients

DETAILED DESCRIPTION:
NLR will be used as predictor for short term survival and patients stay in ICU in 2 groups of patients . Investigators will use it in a group of Medical Critically ill patients as respiratory failure , neuromuscular disorders , renal impairment . the other group is the critically ill surgical patients , as patients with multiple trauma , post major surgery

ELIGIBILITY:
Inclusion Criteria:

* Critically ill trauma patients

Exclusion Criteria:

* auto immune disease endocrine disease renal dysfunction hepatic dysfunction malignancy smoking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 adult patients who are admitted to critical care unit in Assiut university Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
short term survival | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No